CLINICAL TRIAL: NCT03025555
Title: COMPARISON OF PATIENT SATISFACTION AND DIMENSIONAL ACCURACY OF INJECTION MOLDED PEEK AND BRE-FLEX MATERIALS FOR BOUNDED REMOVABLE PARTIAL DENTURES (Randomized Clinical Trial)
Brief Title: Patient Satisfaction and Dimensional Accuracy of Bre Flex and Peek for Removable Partial Dentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sylvia Sami Melek Ekladios, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1987
Record Dates: First submitted 2017-01-12; First posted 2017-01-19 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Patient Satisfaction
Keywords: nylon; polyamide; PEEK; partial denture
MeSH Terms: conditions — Patient Satisfaction | interventions — polyetheretherketone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group 1 (Active Comparator): patients will receive partial denture constructed from breflex material.
  Interventions: Other: Bre.flex
- group 2 (Experimental): patients will receive partial denture constructed from PEEK material.
  Interventions: Other: PEEK

INTERVENTIONS:
Other: PEEK — Polyetheretherketone (PEEK) is a synthetic, tooth colored polymeric material that has been used as a biomaterial in orthopedics for many years but recently used as removable prosthetic material. Advantages of this polymer material are elimination of allergic reactions, high polishing qualities, low plaque affinity, and good wear resistance.
  It has been proven that it shows high mechanical and biological properties. Studies evaluating the properties of this material are limited and need more clinical tests.
  Arms: group 2
Other: Bre.flex — Bre.flex is a nylon-based thermoplastic material, composed of nylon PA 12 (polyamide).Nylon exhibits high physical strength, heat resistance and chemical resistance. It can be easily modified to increase stiffness and wear resistance. Nylon resin can be semi-translucent and provides excellent esthetics but it is a little more difficult to adjust and polish.
  Arms: group 1

SUMMARY:
Evaluation the patient satisfaction and dimensional stability of upper removable partial denture constructed from two different flexible thermoplastic materials.(BRE-FLEX and PEEK).

DETAILED DESCRIPTION:
The assessor is responsible for all clinical procedure that will be conducted in this study during all the visits:

Panoramic radiograph and periapical radiographs will be made on the prospected abutment teeth to evaluate the crown-root ratio, the apical condition of the abutment and their alveolar bone support.

The preliminary impression will be performed with irreversible hydro-colloid impression material (alginate), The impressions will be poured with type IV dental stone to obtain diagnostic casts. Maxillary Face-bow will be recorded. The diagnostic casts will be mounted on semi adjustable articulator in centric occluding relation to evaluate the interarch distance and occlusal plane.

Special trays will be constructed and Mouth preparation will be performed by preparing guiding planes and rests seats will be prepared opposing to the edentulous area. Final impression will be taken by elastomeric impression material. The impression will be poured into type IV dental stone in order to obtain master cast. The master cast will be surveyed. The proposed design will be as follows: metal framework base saddle for edentulous areas on both sides connected with palatal strap. Aker's clasp on all abutments with buccal retention. The denture base will be tried in with acrylic teeth in patient's mouth. After that, the denture base of the partial denture will be processed incorporation with the metal framework into the two different materials to be evaluated. The first group will receive the partial denture in which the metal framework incorporated with the denture base fabricated from PEEK material. The second group will receive the partial denture in which the metal framework incorporated with the denture base material fabricated from BRE-FLEX.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have Kennedy class III modification I upper partially edentulous ridges.
* The remaining teeth have good periodontal condition, with no signs of attrition or gingival recession.
* Male or female patient with age range (45-55) and in good medical condition
* All patients have skeletal Angle's class I maxillo-mandibular relationship and have sufficient interarch distance.
* Free from any systemic or neuromuscular disorder that might affect chewing efficiency of masticatory muscles.
* Free from any tempro-mandibular joint disorder.
* The patients have good oral hygiene and low caries index.

Exclusion Criteria:

* Patients having abnormal habits as bruxism or clenching
* Patients having hormonal disorders as diabetes, thyroid or parathyroid hormonal diseases were not included.
* Teeth with compromised bone support.
* Patient with xerostomia or excessive salivation.
* Patient with abnormal tongue behavior and/or size.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-03-30 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 1 month
  The first week at the time of insertion measuring patient satisfaction immediately after partial denture insertion, The third week measuring patient satisfaction of the partial denture, The fourth week measuring patient satisfaction of the partial denture.
  the patient satisfaction is measured by questionnaire.

SECONDARY OUTCOMES:
dimensional stability | 1 month
  The first week at the time of insertion measuring the dimensional stability immediately after partial denture insertion.
  The third week measuring the dimensional stability of the partial denture,The fourth week measuring the dimensional stability of the partial denture.
  dimensional stability is measured by digital caliper.

IPD SHARING:
Plan to Share IPD: Undecided